CLINICAL TRIAL: NCT01069250
Title: Serial Measurement of Static and Dynamic Cerebrovascular Autoregulation After Brain Injury
Brief Title: Dynamic and Static Autoregulation After Brain Injury
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Patrick Schramm, MD, Johannes Gutenberg University Mainz
Other Study IDs: 2001 448/01
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Acute Brain Injuries; TBI (Traumatic Brain Injury); Intracranial Hemorrhages
Keywords: dynamic cerebrovascular autoregulation; static cerebrovascular autoregulation; acute brain injury; transcranial Doppler ultrasound; critical care
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain injury: Patients after traumatic brain injury or spontaneous intracranial bleeding
  Interventions: Other: There are no interventions in this study

INTERVENTIONS:
Other: There are no interventions in this study

SUMMARY:
The aim of the study assesses static and dynamic cerebrovascular autoregulation daily over one week in patients with traumatic brain injury or intracranial hemorrhage to quantify the temporal profile of the autoregulatory status.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury
* Intracranial hemorrhage

Exclusion Criteria:

* Measurement of TCD were impossible
* Injury of the legs (if the both tigh cuffs for dynamic autoregulation could not be fixed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after traumatic brain injury or intracranial bleeding wich had a Glasgow-Coma-Scale (GCS) of less than 8 and were initially sedated, intubated and mechanically ventilated.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2001-08; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Disturbed cerebrovascular autoregulation after brain injury | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Germany

REFERENCES:
- [Result] Schramm P, Klein KU, Pape M, Berres M, Werner C, Kochs E, Engelhard K. Serial measurement of static and dynamic cerebrovascular autoregulation after brain injury. J Neurosurg Anesthesiol. 2011 Jan;23(1):41-4. doi: 10.1097/ANA.0b013e3181f35854. PMID 21252706